CLINICAL TRIAL: NCT05096390
Title: Multicenter Phase II Study of Axitinib +/- Pembrolizumab in First Line Treatment for Patients With Locally Advanced or Metastatic Papillary Renal Cell Carcinoma (PRCC)
Brief Title: Axitinib +/- Pembrolizumab in First Line Treatment of mPRCC
Acronym: PAXIPEM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAXIPEM (ET21-023); ET21-023 (Other: Centre Leon Berard)
Record Dates: First submitted 2021-10-14; First posted 2021-10-27 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Papillary Renal Cell Carcinoma Type 2
Keywords: PRCC
MeSH Terms: interventions — Axitinib; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, prospective, phase II study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- axitinib + pembrolizumab (Experimental): Axitinib will be administrated orally 5 mg twice a day, with a dose adaptations to the manufacturer recommendations in both groups. Doses can be increased up to 10 mg twice daily.
  Pembrolizumab will be administrated intravenously (IV) over 30 minutes at the dose of 200 mg every 3 weeks according to recent summary of product characteristics (SPC) together with axitinib.
  Interventions: Drug: Axitinib Oral Tablet [Inlyta]; Drug: Pembrolizumab Injection [Keytruda]
- axitinib alone (control) (Active Comparator): Axitinib will be administrated orally 5 mg twice a day, with a dose adaptations to the manufacturer recommendations in both groups. Doses can be increased up to 10 mg twice daily.
  Interventions: Drug: Axitinib Oral Tablet [Inlyta]

INTERVENTIONS:
Drug: Axitinib Oral Tablet [Inlyta] — Axitinib 5 up to 10mg twice a day
Drug: Pembrolizumab Injection [Keytruda] — Pembrolizumab intravenously over 30 min minutes at 200 mg every 3 weeks
  Arms: axitinib + pembrolizumab

SUMMARY:
Multicenter Phase II Study of Axitinib +/- Pembrolizumab in First Line Treatment for Patients With Locally Advanced or Metastatic Papillary Renal Cell Carcinoma (PRCC)

DETAILED DESCRIPTION:
Papillary renal cell carcinoma (PRCC) is the second most common subtype of renal carcinoma accounting for approximatively 10-15% of all renal cancers. Different types of PRCC have been described on the basis of two histologic subtypes, type 1 in 25 to 30% cases, and type 2, with a worse prognosis reported for type 2 metastatic disease. There is currently no standard of care specifically dedicated to metastatic PRCC patients (mPRCC) and treatments developed for metastatic clear cell carcinomas are commonly used ; therefore, mPRCC enrollment in clinical trials is encouraged.

Clinical trials investigated treatments such as sunitinib, or everolimus approved for advanced clear cell carcinoma, or the dual kinase inhibitor directed both towards VEGF receptors (VEGFr) and the MET pathway foretinib, or more recently, the selective MET inhibitor savolitinib. Response rates (RR) were disappointing since generally below 15%, except in a subset of patients with MET germline alterations.

Axitinib which is indicated as second-line treatment in advanced clear cell carcinoma was investigated in a recent specific trial : the Axipap trial. This multicentric phase II trial was conducted after central pathology review to confirm the histologic subtype and a central review was performed to assess the primary endpoint : the 24 week progression free rate (24wPFR). With a median follow up time of 30 months this 24wPFR was found to be over 45%. The best response rate was 28.6% according to the investigators with a median duration of response near 8 months. The investigator assessed response rate was 35.7% in the type 2 subgroup indicating a more important effect of anti-VEGFr in this subtype than in the type 1. The median PFS was around 6 months and was virtually identical in both subtypes.

Recently, some preliminary results of the use of Immune Checkpoint Inhibitors in metastatic non clear cell carcinoma were made available. The PD1 directed antibody Pembrolizumab showed a 28% response rate in 118 patients with papillary tumors including a 6% complete remission rate ; the median duration of response was of 15.3 [2.8-21.0+] months. Atezolizumb (anti-PDL1) combined with Bevacizumab and Durvalumab (anti-PDL1) combined with savolitinib (Met directed TKI) obtained response rates in the same range. These preliminary results demonstrated the potential interest of combining axitinib with an immune check point inhibitor. The results of pembrolizumab as monotherapy were obtained in the largest subset with mPRC.

According to these results obtained, the combination of axitinib and pembrolizumab seems promising in type 2 papillary tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years on the day of signing informed consent.
2. Metastatic or locally advanced (inoperable) type 2 or mixed PRCC, histologically confirmed by central review: FFPE blocks (or all HES and IHC slides) with the initial histology report must be sent for central reading before confirmation of inclusion in the study.
3. No prior systemic treatment for renal cancer (chemotherapy, immunotherapy, anti-angiogenic drugs, or treatment under evaluation) even in adjuvant setting.
4. At least one measurable site of disease according to RECIST v1.1.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤ 1 evaluated within 7 days prior to the date of inclusion.
6. In case of prior radiation therapy, discontinuation of irradiation for at least 3 weeks before first dose of study treatment, with at least 1 site kept/preserved for evaluation. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤ 2 weeks - limited field (<10% of the whole body)) to non-CNS disease.
7. Adequate bone-marrow, hepatic, and renal functions within 14 days prior to the inclusion, with:

   * Hemoglobin ≥ 9.0 g/dl ou ≥ 5.6 mmol/l, neutrophils ≥ 1 000/mm3 (1.0 G/l), Platelets ≥ 100 000/mm3 (100 G/l),
   * Serum creatinine ≤ 2 x ULN OR creatinine clearance ≥ 50 ml/min/1.73m2 (calculated using either MDRD or CKD-EPI formula),
   * AST and ALT ≤ 2.5 x ULN (or ≤ 5 x ULN in case of liver metastasis),
   * Total serum bilirubin ≤ 1.5 x ULN (or direct bilirubin ≤ ULN for participants with total bilirubin levels >1.5 × ULN),
8. Absence of significant proteinuria (<0.5 g/24h) confirmed by urinary dipstick test. If the dipstick test is ≥ 2+, proteinuria will be quantitated on a complete 24h urine sample (< 1 g/l of protein/24h sample)
9. Covered by a medical/health insurance.
10. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
11. Patients of childbearing potential accepting to use effective contraception or abstain from heterosexual activity during study treatment and within 4 months after final dose of study therapy or being surgically sterile. Refer to Appendix 1 for approved methods of contraception.
12. Signed and dated approved informed consent form before any study specific procedures or assessments.

Exclusion Criteria:

1. Presence of brain metastases on Magnetic Resonance Imaging (MRI) or Computed Tomography-scan (CT-scan) performed within 28 days prior to inclusion. Patients with a history of brain metastases treated by surgery or stereotactic surgery, with normal brain MRI or CT-scan are allowed to participate.
2. Metastases with high risk of nervous compression or bone lesion with high risk of fracture.
3. Prior history of other malignancies other than PRCC (except for curatively treated basal cell or squamous cell carcinoma of the skin or in situ uterine cervix carcinoma) unless the subjects has been free of the disease for at least 5 years.
4. Major surgical procedure, open biopsy, or serious none healing wound within 28 days prior to inclusion.
5. Significant cardiovascular disease, including:

   * Disorder of left ventricular function with a left ventricular ejection fraction (LVEF) < 50%,
   * Uncontrolled arterial hypertension under adapted medication: systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 90 mmHg or both despite appropriate therapy, blood pressure must be monitored and controlled before inclusion, or patients under 3 antihypertensive therapies at screening,
   * Myocardial infarction, severe angina, or unstable angina within 6 months prior to inclusion,
   * History of serious ventricular arrhythmia (ie ventricular tachycardia or ventricular fibrillation),
   * Cardiac arrhythmias requiring anti-arrhythmic medications (except for atrial fibrillation that is well controlled with anti-arrhythmic medication),
   * Coronary or peripheral artery bypass graft or active coronary stent within 6 months prior to inclusion,
   * Veinous thrombosis or pulmonary embolism within 6 months prior to inclusion.
6. Any anti-coagulation therapy except prophylactic low dose.
7. History of auto-immune disease except thyroiditis more than 6 months ago.
8. History of any allograft.
9. HIV, HBV, HCV active infections.
10. Any active acute or chronic or uncontrolled infection/disorder that would impair the ability to evaluate the patient or the ability for the patient to complete the study.
11. Known history of active TB (Bacillus Tuberculosis).
12. Interstitial lung disease, respiratory insuffisancy whatever the cause.
13. Prior (non-infectious) pneumonitis requiring systemic corticosteroid therapy or current pneumonitis.
14. Inability to swallow oral medications, or presence of active inflammatory bowel disease, partial or complete bowel obstruction or chronic diarrhea.
15. History of severe hypersensitivity to another monoclonal antibody.
16. Known hypersensitivity to the active substances or to any of the excipients.
17. Receiving or having received immunosuppressive therapy or corticosteroids within 1 month prior to inclusion (except for hydrocortisone for substitution purposes).
18. Live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed. COVID-19 vaccine is allowed if non-living/inactivated.
19. Psychological, familial, sociological, or geographical conditions that would limit compliance with study protocol requirements or known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
20. Inclusion in another clinical trial, except for supportive care trials.
21. Pregnant or breastfeeding woman or patient expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 4 months after the last dose of study treatment (mandatory negative serum or urinary pregnancy test at study entry for all women of childbearing potential).
22. Under or requiring tutorship or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy of axitinib + pembrolizumab versus axitinib in patients with locally advanced or metastatic type 2 papillary renal carcinoma in first-line treatment. | At 6 months for each patient
  6-month objective response rate (6m-ORR), defined as the proportion of patients with CR or PR at 6 months

SECONDARY OUTCOMES:
Duration of response (DOR) | Week 4, 7, 9-10, 18-19, 27-28 then Months 8, 10, 12, 14, 16, 18, 20, 22, 24
  Duration of response in each arm, calculated from the date of first documented response to the date of first documented progression or death.
Best overall response (BOR) using RECIST 1.1 | Up to 24 months for each patient
  Best overall response in each arm, defined as the best response according to RECIST v1.1 recorded from baseline until the end of the study (treatment).
Progression-free survival (PFS) | Up to 24 months for each patient
  PFS in each arm, defined as the time from the date of first treatment administration to the date of documented progression or death from any cause.
Overall survival (OS) | Up to 48 months
  OS in each arm, defined as the time from the date of first treatment administration to the date of death from any cause.
Incidence of adverse events | Up to 48 months
  Safety profile, determined using NCI CTC-AE grading scale v5

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie NEGRIER, PhD, Principal Investigator — Centre Leon Berard
Locations (12):
- France (12):
  - Ico - Paul Papin, Angers
  - CHU de BESANCON, Besançon
  - Chu Bordeaux, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Leon Berard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Centre Antoine Lacassagne, Nice
  - Ap-Hp Hôpital Europeen Georges Pompidou, Paris
  - Ico-Rene Gauducheau, Saint-Herblain
  - Iuct-Oncopole Institut Claudius Regaud, Toulouse
  - Institut de Cancerologie de Lorraine - Alexis Vautrin, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif